CLINICAL TRIAL: NCT07381062
Title: Total Knee Arthroplasty in Conjunction With Intra-operative Genicular Nerve Radio-Frequency Ablation, A Randomized Controlled Clinical Trial
Brief Title: Total Knee Arthroplasty in Conjunction With Intra-operative Genicular Nerve Radio-Frequency Ablation
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ain Shams University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: FMASU MD39/2022
Record Dates: First submitted 2026-01-24; First posted 2026-02-02 (Actual); Last update posted 2026-02-11 (Actual); Status verified 2026-02

CONDITIONS: Post Operative Pain; Functional Outcome
Keywords: Radio-Frequency Ablation; Total Knee Arthroplasty; Genicular nerve; Total knee arthroplasty functional outcome
MeSH Terms: conditions — Pain, Postoperative | interventions — Arthroplasty, Replacement, Knee

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control (Active Comparator): underwent Total knee arthroplasty only
  Interventions: Procedure: Total knee arthroplasty
- Genicular nerve radio-frequency ablation (Experimental): underwent Total knee arthroplasty with genicular nerve radio-frequency ablation
  Interventions: Procedure: Total knee arthroplasty; Procedure: Genicular nerve radiofrequency ablation

INTERVENTIONS:
Procedure: Total knee arthroplasty — Conventional Total knee arthroplasty operation performed
  Other Names: knee joint replacement
Procedure: Genicular nerve radiofrequency ablation — Genicular nerve radiofrequency ablation done with no modifications except being performed with total knee arthroplasty in the same setting
  Arms: Genicular nerve radio-frequency ablation

SUMMARY:
The aim of this study is to compare between conventional Total Knee Arthroplasty (TKA) and Total Knee Arthroplasty (TKA) combined with intra-operative Genicular Nerve Radio-Frequency Ablation (GNRFA), concerning post-operative functional outcome and pain scores in patients with advanced knee osteoarthritis

DETAILED DESCRIPTION:
The aim of this study is to compare between conventional Total Knee Arthroplasty (TKA) and Total Knee Arthroplasty (TKA) combined with intra-operative Genicular Nerve Radio-Frequency Ablation (GNRFA), concerning post-operative functional outcome and pain scores in patients with advanced knee osteoarthritis

Including 70 knees randomized using a computer-generated sequence into two groups, the first group underwent TKA combined with GNRFA, and the other group underwent TKA only. All the TKA surgeries were performed by a single surgeon including patients aged from fifty to eighty years with advanced primary knee osteoarthritis from both sexes

ELIGIBILITY:
Inclusion Criteria:

* Patients with advanced knee osteoarthritis
* Both sexes
* Age from 50-80 years old

Exclusion Criteria:

* Patients underwent previous GNRFA
* Patients underwent previous knee surgery
* patients requiring constrained knee arthroplasty prosthesis (with extreme deformities)

Ages: 50 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 70 (Actual)
Dates: Start 2022-02-22 (Actual); Primary Completion 2024-03-04 (Actual); Study Completion 2024-10-01 (Actual)

PRIMARY OUTCOMES:
Post operative pain | 6 months post operative
  pain assessment using Visual analogue scale, minimum value is 0 meaning no pain and maximum value is 10 meaning the worst pain, higher score means worse outcome
Post operative knee functional outcome | 6 months
  measuring the knee functional outcome post operative using oxford knee score, minimum score is 0 meaning the worse outcome and maximum is 48 meaning the best outcome. higher score means better outcome

CONTACTS AND LOCATIONS:
Overall Officials: Assem Mohamed Mahmoud Ahmed, MD, Principal Investigator — Ain Shams University
Locations (1):
- Ain Shams University, Cairo, Abbassia, Egypt

IPD SHARING:
Plan to Share IPD: Undecided
No need to contact them

DOCUMENTS (1):
  • Study Protocol (2022-01-12): https://cdn.clinicaltrials.gov/large-docs/62/NCT07381062/Prot_001.pdf